CLINICAL TRIAL: NCT04103710
Title: Prevalence of Molar Incisor Hypo Mineralization Among Children Who Have Been Treated With Asthmatic Drugs During Their First Three Years of Life(A Cross- Sectional Study)
Brief Title: Prevalence of Molar Incisor Hypomineralization Among Children Treated With Asthmatic Drugs Early in Their Lives
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marina Girgis Azmy, dentist, Cairo University
Other Study IDs: MIH and asthmatic children
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Molar Incisor Hypomineralization; Asthma in Children
Keywords: MIH; asthmatic drugs
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the prevalence of molar incisor hypo mineralization among children who have been treated with asthmatic drugs during the first three years of life.

DETAILED DESCRIPTION:
The term Molar incisor hypo mineralization (MIH) was first introduced in 2001 as a developmental disorder of enamel characterized by hypo mineralization -of systemic origin - affecting the enamel of first permanent molars (PFM) ,frequently associated with affected permanent incisors.

The prevalence of MIH varies widely, ranging from 2.4 % to 40.2% in different populations. This wide variation may be due to differences in diagnostic criteria and methodologies used by the authors. Concerning the etiology of MIH it is mostly related to pre natal, perinatal, and post natal illness.

Asthma and asthmatic drugs have been proposed to be one of the etiological factors of MIH,Internationally, the mean prevalence of pediatric asthma is 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Children from 8 to 12 years old with fully erupted first permanent molars and permanent incisors.
2. Children who were patients of the Pediatric Pulmonary Clinic and had used asthma drugs (oral and inhaled bronchodilators or corticosteroids) during their first three years of life.

Exclusion Criteria:

1. Children with any chronic disease
2. Children with unerupted or partially erupted first permanent molars.
3. Children using a fixed orthodontic appliance
4. Children having extensive carious lesions that might mask dental enamel defects.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged from 8 to 12 years old with fully erupted first permanent molar and permanent incisors, who have been treated with any type of asthmatic drugs during their first three years of life.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of molar incisor hypo mineralization (MIH) | baseline
  - Clinical examination will be carried out by the principle investigator using mirror and probe to examine all surfaces of each first permanent molar &permanent incisors following the diagnostic criteria of MIH set by the European Academy of Pediatric Dentistry (EAPD)as following :Demarcated opacities:
  Enamel disintegration:
  Atypical restorations:
  Extracted teeth:
  Tooth sensitivity:

SECONDARY OUTCOMES:
the severity of MIH | baseline
  the severity of MIH will be recorded into three categories :Mild MIH , Moderate MIH, and Severe MIH

CONTACTS AND LOCATIONS:
Overall Officials: Marina G Azmy, BSc., Principal Investigator — BSc.Faculty of Dentistry, Cairo University, 2012; Marwa A Foad, MSc, Study Chair — Lecturer of Pediatric Dentistry and Dental Health; soad Abd el Moneam, PhD, Study Director — Associate Professor of Pediatric Dentistry and Dental Public Health
Locations (1):
- Agouza police hospital, Giza, Egypt

REFERENCES:
- [Background] Loli D, Costacurta M, Maturo P, Docimo R. Correlation between aerosol therapy in early childhood and Molar Incisor Hypomineralisation. Eur J Paediatr Dent. 2015 Mar;16(1):73-7. PMID 25793958
- [Background] Wogelius P, Haubek D, Nechifor A, Norgaard M, Tvedebrink T, Poulsen S. Association between use of asthma drugs and prevalence of demarcated opacities in permanent first molars in 6-to-8-year-old Danish children. Community Dent Oral Epidemiol. 2010 Apr;38(2):145-51. doi: 10.1111/j.1600-0528.2009.00510.x. Epub 2010 Jan 4. PMID 20059490
- [Background] Visweswar VK, Amarlal D, Veerabahu R. Prevalence of developmental defects of enamel in children and adolescents with asthma: a cross-sectional study. Indian J Dent Res. 2012 Sep-Oct;23(5):697-8. doi: 10.4103/0970-9290.107432. PMID 23422632
- [Background] Guergolette RP, Dezan CC, Frossard WT, Ferreira FB, Cerci Neto A, Fernandes KB. Prevalence of developmental defects of enamel in children and adolescents with asthma. J Bras Pneumol. 2009 Apr;35(4):295-300. doi: 10.1590/s1806-37132009000400002. English, Portuguese. PMID 19466266
- [Background] Mastora A, Vadiakas G, Agouropoulos A, Gartagani-Panagiotopoulou P, Gemou Engesaeth V. Developmental defects of enamel in first permanent molars associated with use of asthma drugs in preschool aged children: A retrospective case-control study. Eur Arch Paediatr Dent. 2017 Apr;18(2):105-111. doi: 10.1007/s40368-017-0280-1. Epub 2017 Mar 2. PMID 28255932